CLINICAL TRIAL: NCT07069881
Title: A Randomized Controlled Trial of Endodontic Treatment Using Sonic-activated Irrigation and Passive Ultrasonic Irrigation to Evaluate Healing in Chronic Apical Periodontitis
Brief Title: Sonic vs Passive Ultrasonic Irrigation for Chronic Apical Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2024-435
Record Dates: First submitted 2025-06-22; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Apical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonic-Activated Irrigation (Experimental)
  Interventions: Device: Sonic-Activated Irrigation
- Passive Ultrasonic Irrigation (Active Comparator)
  Interventions: Device: Passive Ultrasonic Irrigation

INTERVENTIONS:
Device: Sonic-Activated Irrigation — Sonic-activated irrigation was performed using the polymer tip (Eddy™, VDW, Germany) activated by an airscaler handpiece.
  Arms: Sonic-Activated Irrigation
Device: Passive Ultrasonic Irrigation — Passive ultrasonic irrigation was performed using the ultrasonic tip (ACTEON, France) attached to an ultrasonic device (P5 Newton™, ACTEON, France)
  Arms: Passive Ultrasonic Irrigation

SUMMARY:
This randomized, controlled, double-blinded clinical trial aims to directly compare the efficacy of Sonically Activated Irrigation (SAI) versus Passive Ultrasonic Irrigation (PUI) in the root canal treatment of teeth with chronic apical periodontitis, analyze potential influencing factors, and thereby identify a highly effective and safe root canal irrigation protocol. The ultimate goal is to provide an evidence-based rationale for optimizing irrigation technique selection and overall treatment strategies for chronic apical periodontitis.

DETAILED DESCRIPTION:
Root canal therapy (RCT) is the common treatment for chronic apical periodontitis. Successful outcomes critically depend on the complete eradication of infection within the root canal system. The efficacy of infection control is significantly influenced by the irrigation technique employed. While passive ultrasonic irrigation (PUI) is a widely utilized form of activated irrigation in clinical practice, it carries inherent risks such as instrument separation and unnecessary dentin removal, limiting its use.

Sonically activated irrigation (SAI) represents a novel irrigation approach. Its polymeric tips circumvent the drawbacks associated with ultrasonic metal tips while delivering comparable irrigation efficiency. However, high-quality randomized controlled clinical evidence supporting its use is currently lacking.

This randomized, controlled, double-blinded clinical trial aims to directly compare the efficacy of SAI versus PUI in root canal treatment of teeth with chronic apical periodontitis and analyze potential influencing factors. The goal is to identify a highly effective and safe root canal irrigation protocol, ultimately providing an evidence-based rationale for optimizing irrigation technique selection and overall treatment strategies for chronic apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate in this study and provide informed consent;
2. Age 18-59 years at the time of enrolment;
3. At least one permanent tooth diagnosed with chronic periapical periodontitis at root development stage of Nolla10th;
4. Able to follow up on schedule.

Exclusion Criteria:

1. Allergies to any medications or materials necessary to complete the procedures;
2. Non-restorable teeth, teeth with severe defects, or teeth that need to be extracted due to orthodontic treatment;
3. Teeth with root canal treatment or vital pulp therapy;
4. Teeth with canal calcification or root canal instrument separation;
5. Teeth with root fracture or vertical root fracture;
6. Tooth with internal or external root resorption;
7. Patients with periodontitis;
8. Patients with orthodontic treatment;
9. Presence of dental phobia;
10. Women who are pregnant;
11. Patients who have taken medications that affect central nervous system, such as tricyclic antidepressant;
12. Patients who have taken medications that affect immune response, such as glucocorticoid or cyclosporin;
13. Patients after radiotherapy of tumor head and neck;
14. Patients who have taken medications that affect curative effect, such as bisphosphonates;
15. Patients with serious systemic diseases that can affect curative effect;
16. Participation in other clinical studies within the past several weeks;
17. Patients who are deemed unsuitable to participate in the study by investigators.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic Effect Evaluation | 12 months after treatment
  1. Success: A tooth is considered successfully treated when it is asymptomatic, showing no signs of apical infection such as percussion pain, mobility (loosening), tenderness, mucosal swelling, sinus tract, or fistula. Radiographically, the periapical radiolucency must demonstrate either absence or significant reduction.
  2. Failure: Treatment is deemed unsuccessful if the tooth remains symptomatic or develops new symptoms of apical infection (e.g., pain, fistula). Radiographically, the size of the periapical radiolucency remains unchanged or shows enlargement.

SECONDARY OUTCOMES:
postoperative pain | day 1 after treatment
  Postoperative pain was assessed using the Visual Analogue Scale (VAS) during clinical follow-up on day 1 after treatment.
Cone Beam Computed Tomography Periapical Index Scores (CBCTPAI) | 12 months after treatment
  The CBCT Periapical Index (CBCTPAI) assigns scores to lesions of chronic apical periodontitis based on the largest dimension measured in three planes (buccopalatal, mesiodistal, diagonal) on CBCT scans.
  0： Intact periapical bone structures；
  1. Diameter of periapical radiolucency > 0.5-1 mm；
  2. Diameter of periapical radiolucency > 1-2 mm；
  3. Diameter of periapical radiolucency > 2-4 mm；
  4. Diameter of periapical radiolucency > 4-8 mm；
  5. Diameter of periapical radiolucency > 8 mm； Score (n) + E： Expansion of periapical cortical bone； Score (n) + D ： Destruction of periapical cortical bone.
The size of the periapical lesion | 12 months after treatment
  The size in periapical lesions were quantified using cone beam computed tomography (CBCT) at 1-year postoperative compared to preoperative baseline across three anatomical planes: buccopalatal, mesiodistal, and diagonal.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Hospital, Southern Medical University, Guangzhou, Guangdong, China